CLINICAL TRIAL: NCT01189916
Title: Transrectal - Natural Orifice Translumenal Endoscopic Surgery (NOTES)
Brief Title: Transrectal NOTES Appendectomy - Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Natural Orifice Surgery Consortium for Assessment and Research (Other)
Responsible Party: Principal Investigator, Anne-Marie Boller, Assistant Professor of Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00023311
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Appendectomy, Laparoscopic; Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transrectal NOTES appendectomy (Experimental): These patients will undergo an experimental surgical procedure that uses flexible endoscopic instruments (i.e., inserted through the rectum).
  Interventions: Procedure: Endoscopically assisted Appendectomy Surgery

INTERVENTIONS:
Procedure: Endoscopically assisted Appendectomy Surgery — Using endoscopic instruments a small incision will be made in the rectum wall and the endoscope will be advanced into the insufflated peritoneal cavity. At least one laparoscopic trocars will be placed through the abdominal wall for laparoscopic instrument insertion to manipulate and cut tissue. The flexible endoscope will provide visualization of the surgical field and flexible endoscopic instruments may be used to augment surgical manipulation with the laparoscopic instruments. The appendix will be removed through the anus. Endoscopic clips, sutures or tissue anchors (TAS)will be used to close the rectal access site.
  Other Names: NOTES; Natural orifice translumenal endoscopic surgery; Transrectal Appendectomy

SUMMARY:
Natural orifice translumenal endoscopic surgery (NOTES) has revolutionized the concept of minimally invasive surgery. NOTES is currently performed through transgastric or transvaginal approaches. The transvaginal approach is technically easier, but is only available to women. A transrectal approach has been proposed as a potential alternative to transvaginal NOTES for men. Fortunately, the technology to facilitate transrectal access and closure for NOTES has been in use for over twenty years, in the form of transanal endoscopic microsurgery (TEM) platforms.

We hypothesize that transrectal NOTES appendectomy is feasible in humans using a flexible endoscope and a TEM platform to assist with transrectal access and closure. After a pre-clinical study involving 5 cadavers, we will perform a clinical study of 10 transrectal NOTES appendectomies in patients already scheduled to undergo laparoscopic total proctocolectomy or total abdominal colectomy. The tissues involved in the NOTES procedure will be removed as part of the patient's originally scheduled operation, reducing the risk of morbidity as a result of an inadequate transrectal closure or appendiceal stump leak. We will measure operative times, complication rates, peritoneal contamination, and assess the integrity of the rectotomy closures. We hope to show that transrectal NOTES appendectomy is clinically feasible in humans using a TEM platform.

DETAILED DESCRIPTION:
Pre-clinical phase: We conducted the first phase of the study in cadavers to troubleshoot the procedures, and to determine the optimal transrectal approach (anterior versus posterior). We have determined the anterior transrectal approach to be feasible and preferable to a posterior transrectal approach.

Clinical phase: The second phase of the project will be a feasibility study involving 10 human patients. We will recruit patients who are already scheduled to undergo elective laparoscopic total proctocolectomy, total abdominal colectomy, completion proctectomy , or sigmoidectomy from the surgical clinics.

Operative procedure: Patients will undergo a standard preoperative mechanical bowel prep, and will receive standard perioperative antibiotics and deep venous thrombosis (DVT) prophylaxis to reduce the risk of surgical site infection and thromboembolic complications, respectively. The subjects will be placed in lithotomy position, and undergo general anesthesia per usual routine. A laparoscopic team and a NOTES team will carry out the operation. The laparoscopic team will obtain laparoscopic access using standard laparoscopic technique. The NOTES team will perform rigid proctoscopy to assess the suitability of the rectum. The Karl-Storz (Tuttlingen, Germany) operating rectoscope will be used for TEM. After positioning the rectoscope, an intraluminal tissue oximetry measurement will be taken at the intended rectotomy site using an FDA-approved endoscopic tissue oximetry probe (T-Stat®, Spectros, Portola Valley, CA) passed through the TEM device. In human patients, we will collect peritoneal fluid for quantitative cultures at two time-points (immediately after peritoneal access, and after rectotomy closure), using a sterile suction trap attached in-line to a laparoscopic suction irrigator to determine the level of contamination from the procedure. The NOTES appendectomy will be completed using the flexible endoscope with laparoscopic assistance as needed. We will remove the specimen through the anus and close the rectal access site with a standard TEM closure. We will then perform a standard intraoperative insufflation test by submerging the pelvis and rectotomy site under saline, and insufflating the rectum to look for bubbles from the rectal closure site. At the conclusion of the NOTES procedures, we will remove the TEM device, and a laparoscopic team will proceed with laparoscopic proctocolectomy or total abdominal colectomy as originally planned. Once the specimen has been removed, we will use a bench-top test to determine the burst-pressure strength of the rectotomy closures. The specimen will be sent to pathology per standard routine, and postoperative care for the proctocolectomy or total abdominal colectomy patients will proceed per usual routine.

Outcome measurements: We will measure operative times, intraoperative complication rates, tissue oxygen saturation at the closure site, and rectotomy closure strength using an intraoperative insufflation test and an ex-vivo burst-pressure test. In the human cases we will also obtain intraoperative quantitative peritoneal fluid cultures to quantify the amount of peritoneal contamination as a result of the NOTES procedures.

Patients will be followed while in the hospital to assess for complications potentially related to the NOTES procedure. They will then return and be evaluated by their surgeon two weeks following their procedure. At this visit, any additional post-operative complications potentially related to the NOTES procedure will be noted in the patient's medical record.

Potential risks of this study include the usual risks involved in a standard laparoscopic proctocolectomy or total abdominal colectomy procedures including bleeding, infection, injury to surrounding structures, port/trocar site pain, anastomotic leak, incontinence, and sexual dysfunction. Additional potential risks include those related to flexible endoscopy, including bowel perforation and bleeding. In addition, there is the possibility that there may be new, unanticipated complications from this modified surgical technique. We estimate that the additional NOTES procedure will add 90 minutes to the general anesthesia time required for the patient's laparoscopic total proctocolectomy. Patient risks will be mitigated by having the procedure performed by surgeons with expertise in advanced laparoscopic, colorectal and NOTES surgery.

This feasibility study will evaluate the potential feasibility of this modified NOTES technique in 10 patients. Once a standardized technique is established and risks are shown to be low, a prospective comparative evaluation is planned to compare this modified approach to other NOTES approaches.

ELIGIBILITY:
Inclusion Criteria:

* ability to undergo general anesthesia
* Age > 18 yrs
* ability to give informed consent
* requires total proctocolectomy,total abdominal colectomy, completion proctectomy, or sigmoidectomy
* absence of exclusion criteria

Exclusion Criteria:

* age < 18
* pregnancy
* emergency operation
* contraindication for laparoscopic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
operative time | intraoperative

SECONDARY OUTCOMES:
perioperative complications | two weeks
closure strength | intraoperative
  Rectotomy closure strength will be measured intraoperatively using air insufflation, as well as postoperatively using pressurized fluid on the specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Boller, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States